CLINICAL TRIAL: NCT05933525
Title: A Randomized, Double-blind, Placebo-controlled Trial Assessing the Efficacy of IMM-124E (Travelan®) in a Controlled Human Infection Model for Enterotoxigenic Escherichia Coli (ETEC)
Brief Title: Clinical Study to Assess the Efficacy of IMM-124E (Travelan®) in a Controlled Human Infection Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immuron Ltd. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMM-124E-002
Record Dates: First submitted 2023-05-26; First posted 2023-07-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diarrhea; Travelers Diarrhea; Infectious Diarrhea
Keywords: Enterotoxigenic E.coli; Travelers diarrhea; prophylactic; ETEC; IMM-124E; Travelan
MeSH Terms: conditions — Diarrhea; Dysentery

STUDY DESIGN:
Intervention Model Description: 60 healthy volunteer participants will be randomized to receive Travelan investigational product or placebo. The study is a double-blind randomized study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Consenting, eligible participants will be randomized in a 1:1 ratio to receive either the test article Travelan® or placebo. Once enrolled into the study (subject meets all eligibility criteria and is selected by the investigator for inclusion in the study), subjects will be assigned a randomization number. The subject will receive the study treatment regimen assigned to the corresponding randomization number. Subjects will receive the test article/placebo in containers bearing their assigned identification numbers. This number will be linked to the randomization code list securely maintained throughout the clinical phase of the study by the designated study staff. Investigators and participants will remain blinded to group assignments until completion of the clinical phase of the trial and validation of the clinical and immunological data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Travelan (Active Comparator): IMM-124E (Travelan) is the investigational product. Travelan 1200mg will be taken orally for 7 days.
  Interventions: Biological: Travelan
- Placebo (Placebo Comparator): ProMilk 85 milk powder is the placebo. Placebo has been manufactured into tablets using the same manufacturing process as Travelan. 1200mg will be taken orally for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Travelan — 6 Travelan tablets (1200mg) administered orally for 7 days
  Other Names: IMM-124E
  Arms: Travelan
Other: Placebo — 6 tablets of placebo (1200mg) administered orally for 7 days
  Other Names: ProMilk 85 milk powder
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to investigate if Travelan® protects healthy adult volunteers from moderate-to-severe diarrhea upon challenge with Enterotoxigenic Escherichia coli (ETEC) strain H10407.

DETAILED DESCRIPTION:
Up to 60 subjects will be randomized to receive either the Travelan® product or a placebo followed by challenge with ETEC strain H10407. Subjects will receive Travelan® or placebo caplets beginning 2 days prior to experimental challenge with ETEC strain H10407. Travelan®/placebo will be administered for a total of 7 days, or until antibiotic treatment has been initiated. Antibiotic treatment will be initiated after early antibiotic treatment criteria are met or 5 days after challenge.

Early antibiotic treatment will commence when any of the following criteria are met and a physician determines it to be warranted:

1. Severe diarrhea based on volume (800 g in 24 hours)
2. Diarrhea of any severity AND 2 or more of the following symptoms: severe abdominal pain, severe abdominal cramps, severe nausea, severe headache, severe myalgias, severe arthralgia), any fever (≥ 38.0°C), or any vomiting
3. Any fever ≥ 39.0°C
4. Subjects who experience unexpectedly severe events such as symptomatic hypotension (disproportionate to volume loss), renal dysfunction, or altered mental state at the discretion of the investigators.
5. A study physician determines that early treatment is warranted for other reasons.

The placebo is a commercially-sourced high-protein milk product repackaged and masked to mirror the Travelan® product.

Upon admission to the inpatient unit, clinical monitoring will consist of daily medical assessments with adverse event (AE) determination, vital signs at least three times daily, examination and weighing of all stools, stool culture work-up for the challenge strain up to three times daily, and safety laboratory tests. Any subject passing a grade 3-5 stool will be encouraged to start drinking oral fluids at a rate equal to 1.5 times their stool output (or at the same rate as their emesis output as applicable). Intravenous (IV) rehydration will be provided if pre-specified criteria are met.

All subjects will be treated with ciprofloxacin (500 mg by mouth twice daily for three days) or other antibiotic where applicable starting five days after ingesting the H10407 challenge inoculum unless early treatment criteria are met. Subjects will be discharged from the inpatient facility when clinical symptoms are resolved or resolving and two consecutive stool cultures (taken at least 12 hours apart) are negative for the ETEC challenge strain. Subjects may be discharged earlier than Day 8 if they meet criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years of age, inclusive at time of screening visit.
2. General good health, without significant medical illness, abnormal vital signs or physical examination findings, or clinical laboratory abnormalities, as determined by the principal investigator (PI) in consultation with the Medical Monitor and Sponsor.
3. Demonstrate comprehension of the protocol procedures, requirements, and CHIM this will be evaluated by completing a multiple choice comprehension assessment (passing grade > 70%) during screening and in the consenting process.
4. Willing to participate, as evidenced by signing the informed consent document.
5. Available for all planned follow-up visits.
6. Negative serum pregnancy test at screening and negative serum and/or urine pregnancy test on the day of admittance to the inpatient unit for all female participants. All females must agree to use an efficacious hormonal or barrier method of birth control during the study. Efficacious methods of birth control include hormonal birth control methods (oral contraceptive pills, patches, vaginal rings, long-acting reversible contraception, surgical sterilization, condoms with spermicide, or abstinence from intercourse with a male partner. Female participants unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).
7. A negative Covid-19 PCR test is required on the day of admission to the unit to comply with Pharmaron's Covid-19 policy (subjects reporting to admission for Cohort 1 who test positive for COVID-19 may rescreen for Cohort 2)
8. Acceptable hematology and blood chemistry levels as assessed by the PI. i.e., Serum creatinine <1.3 mg/dL. AST, GGT, amylase, lipase, alkaline phosphatase not to exceed 1.5x upper limit of normal (ULN)
9. Vital signs will be assessed in the supine position and must be within the following ranges:

   * Oral body temperature between 35-37oC inclusive
   * Systolic blood pressure between 90-140 mmHg inclusive
   * Diastolic blood pressure between 55-90 mmHg inclusive
   * Pulse rate between 45-90 bpm inclusive

Exclusion Criteria:

1. Presence of a significant medical condition (e.g., psychiatric conditions such as significant anxiety, depression, or somatization disorder; gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis/dyspepsia, gastroesophageal reflux disease, inflammatory bowel disease, or irritable bowel syndrome (as suggested by medical history or medical diagnosis); history of major gastrointestinal surgery; or laboratory abnormalities that in the opinion of the investigator preclude participation in the study. Significant medical conditions include HIV, active Hepatitis B or C infection, ongoing immunosuppression for any reason, autoimmune disease, any underlying cardiac, pulmonary, endocrine, or renal conditions, any gastrointestinal illness (chronic reflux, inflammatory bowel disease, ulcer), any diabetes mellitus, and other such illnesses that can put a volunteer at increased risk. Exclusionary laboratory abnormalities include any abnormality that is grade 2 or above, or any two grade 1 laboratory abnormalities.
2. Immunosuppressive illness or evidence of IgA deficiency (serum IgA levels outside the normal range). This includes any disease that requires immunosuppressive medication such corticosteroids, monoclonal antibodies that target key aspects of the immune system (e.g. rituximab or TNF-blockers, or any autoimmune disease).
3. Positive serology results for HIV, HBsAg, or HCV antibodies, and confirmatory tests if appropriate.
4. Positive urine drug screen (positive for the presence of amphetamines, barbiturates, opiates, phencyclidine, cocaine, benzodiazepines, methadone, and propoxyphene at screening and at the discretion of the study physician, with the exception of stable persons with a diagnosis of ADHD that is well-controlled with a prescribed amphetamine.
5. History of alcohol abuse in the past 3 months or drug abuse in the past year
6. Significant abnormalities in screening laboratory hematology, serum chemistry or electrocardiogram, as determined by the PI or PI in consultation with the Medical Monitor and Sponsor. Significant ECG abnormalities include the following:

   1. PR > 220 msec
   2. QRS complex > 120 msec
   3. QTcF > 450 msec (male) or >460 msec (female)
7. Serum bilirubin exceeds upper limit of normal
8. Use of any medication known to affect immune function (e.g., corticosteroids and others) within 30 days preceding receipt of the investigational products or planned to be used during the active study period. Any regular systemic corticosteroid will be exclusionary, while topical, intranasal, and inhaled steroids will be permitted.
9. Nursing or lactating on the day of admittance to the inpatient unit.
10. Inability to tolerate 150 ml of sodium bicarbonate buffer.
11. Recent vaccination (including licensed vaccines) or receipt of an investigational product (within 30 days before challenge through 30 days following the challenge dose).
12. History of diarrhea (> 3 unformed or liquid stools over a 24-hour period) in the 2 weeks prior to the planned inpatient phase.
13. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency, or loose or liquid stools other than on an occasional basis.
14. Regular use of laxatives or any agent that increases gastric pH (regular defined as at least weekly).
15. Use of proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
16. A fever (≥38.0°C) in the 2 weeks prior to time of challenge.
17. Use of antibiotics during the 30 days before bacterial dosing or receipt of more than 3 courses of antibiotics over the two months prior to dosing.
18. Blood or plasma donation of one pint or more within 30 days preceding the receipt of the investigational products.
19. Lactose intolerance or allergy to milk or milk products.
20. Employment as a health care worker, food handler, childcare worker, or caregivers for elderly or immunocompromised individuals.
21. Allergy to fluoroquinolones, trimethoprim-sulfamethoxazole, doxycycline, or ampicillin/penicillin (excluded if allergic to two of four).
22. History of microbiologically confirmed ETEC infection in the last 3 years.
23. Occupation involving handling of ETEC currently, or in the past 3 years.
24. Symptoms consistent with travelers' diarrhea defined as >3 unformed or liquid stools over a 24 hour period concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study. ETEC endemic countries include all countries in Asia (except for Japan and South Korea) the Middle East, Africa, Mexico, Central and South America.
25. Vaccination for or ingestion of ETEC, cholera, Shigella, or E. coli heat-labile toxin within 5 years prior to dosing.
26. Any prior experimental infection with ETEC strain H10407, or prior experimental infection with other ETEC strains or other bacterial enteric pathogens (Salmonella, Shigella, and Campylobacter) within the past 5 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To measure the protective efficacy of oral administration of Travelan compared to placebo against moderate-to-severe diarrhea following with E.coli (ETEC) challenge. | Monitoring for the Inpatient Study Phase, Study Days -3 to Day 8 or day of dismissal from the clinical trial facility
  The number of subjects who encounter moderate to severe diarrhea (defined as ≥4 Grade 3-5 stools in any 24-hour period post-challenge or ≥401 grams of Grade 3-5 stools in any 24-hour period post-challenge) will be recorded for the Travelan group and the placebo group.
  All stool samples will be collected, weighed and graded.
  Stool grading scale:
  Grade 1 = Fully formed (normal) Grade 2 = Soft (normal) Grade 3 = Thick liquid (diarrheal) Grade 4 = Opaque watery (diarrheal) Grade 5 = Rice-water (diarrheal).
  Diarrhea (Grade 3-5 stools) severity in a 24 hour period (1g = 1ml):
  1-mild (2-3 loose/liquid stool totaling <400 g), 2-moderate (4 to 5 loose/liquid stools or >401 to 800 g), 3-severe (6 or more loose/liquid stools totaling >800 g).

SECONDARY OUTCOMES:
Subjects requiring oral rehydration solution and/or intravenous fluids post ETEC challenge for the Travelan group and the placebo group | Monitoring post challenge on Study Days 1-8 or Day of dismissal from the clinical trial facility.
  Measurement of the number of subjects who require oral rehydration solution and/or intravenous fluids on one or more days post challenge. Numbers will be monitored daily and expressed as a percentage of the Travelan or placebo group.
Density of ETEC organisms in post-challenge stool samples at 48 hours post ETEC challenge for the Travelan group and the placebo group | Monitoring on Study Day 3 or 48 hours post challenge
  The number of colony forming units (CFUs) of ETEC challenge strain measured by quantitative bacterial stool culture 48 hours post challenge per gram of stool (1g = 1ml).
Safety and tolerability of oral doses of Travelan compared to placebo. Measurement ofthe number of AEs graded as moderate-to-severe (Grade 2-4) for Diarrhea, fever, vomiting and other listed AEs as assessed using the CTCAE v5.0 criteria for AEs. | Monitoring for the inpatient study phase: Study Days -3 to Day 8 or day of dismissal from the clinical trial facility.]
  All AEs will be recorded for the Travelan group and the placebo group using the following criteria (1-4):
  1. Diarrhea severity (Grade 3-5 stools) in a 24 hour period (1g = 1ml):1-mild (2-3 loose/liquid stool totaling <400 g), 2-moderate (4 to 5 loose/liquid stools or >401 to 800 g), 3-severe (6 or more loose/liquid stools totaling >800 g).
  2. Temperature maximum measured in a 24 hr period: no fever (<38.0°C), 1-mild (38.0-38.4°C), 2-moderate (38.5-38.9°C), 3-severe (>39.0°C); 4-Potentially life threatening (>40oC).
  3. Vomiting in a 24 hr period: 0-no episodes, 1-mild (1-2 episodes), 2-moderate (2-3 episodes), or 3-severe (>5 episodes).
  4. Nausea, abdominal discomfort and pain, abdominal cramps, headache, malaise or anorexia graded as follows: 0-Non-existent, 1 -mild (not interfering with routine activities), 2 -moderate (interfering but not precluding routine activities), 3 -severe (precluding routine activities), 4 - potentially life threatening (requires hospitalization)
Percent of subjects with severe diarrhea post ETEC challenge for the Travelan group and the placebo group | Monitoring post challenge on Study Days 1-8 or Day of dismissal from the clinical trial facility.
  Severe diarrhea defined as 6 or more loose liquid stools in a 24 hour period totaling >800g. (1g = 1ml).
  All stools will be collected, weighed (1g = 1ml) and graded.
  Stool Grading Scale:
  Grade 1 = Fully formed (normal) Grade 2 = Soft (normal) Grade 3 = Thick liquid (diarrheal) Grade 4 = Opaque watery (diarrheal) Grade 5 = Rice-water (diarrheal).
  Diarrhea severity (Grade 3-5 stools) in a 24 hour period post-challenge (1g = 1ml):
  1-mild (2-3 loose/liquid stool totaling <400 g), 2-moderate (4 to 5 loose/liquid stools or >401 to 800 g), 3-severe (6 or more loose/liquid stools totaling >800 g).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MB,ChB,FACP, Principal Investigator — Pharmaron Clinical Pharmacology Center
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No